CLINICAL TRIAL: NCT05220254
Title: Stanford Tobacco Treatment Services - Virtual Reality Treatment for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Judith Prochaska, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-60253; P30CA124435 (NIH)
Record Dates: First submitted 2021-12-13; First posted 2022-02-02 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; MindCotine Virtual Reality Mindful Exposure Therapy
Keywords: Virtual Reality; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MindCotine mobile app program (Experimental)
  Interventions: Behavioral: MindCotine's VR app

INTERVENTIONS:
Behavioral: MindCotine's VR app — The MindCotine program would be a 6-week intervention to help users utilize mindfulness based skills, and involves virtual exposure therapy.

SUMMARY:
This study aims to see how feasible a mobile app based virtual reality program for smoking cessation (MindCotine) would be among Stanford cancer center patients

ELIGIBILITY:
Inclusion Criteria:

* Daily cigarette smoker or some day smoker (>9 cigarettes per week)
* Age 18+
* English or Spanish fluent
* Smartphone compatibility
* Available to interact with a smartphone app for 6-weeks
* Available to complete the EOT assessment at end of 6-weeks
* Ability to understand and the willingness to personally sign the written IRB-approved informed consent document.
* Confirm phone, email, address during consent

Exclusion Criteria:

* Ever had epilepsy
* Less than 10 cigarettes per week
* Not English or Spanish fluent
* No smartphone compatibility
* Unavailable to interact with the VR program,
* Unavailable to answer questions about the intervention post-treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson RW, Cao-Nasalga A, Chieng A, Pirkl A, Jagielo AD, Xu C, Goldenhersch E, Rosencovich N, Waitman C, Prochaska JJ. Adding Virtual Reality Mindful Exposure Therapy to a Cancer Center's Tobacco Treatment Offerings: Feasibility and Acceptability Single-Group Pilot Study. JMIR Form Res. 2024 Jul 23;8:e54817. doi: 10.2196/54817. PMID 39042439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants use the app for 6 weeks and complete a final end of treatment survey.
Pre-assignment Details: 105 participants were screened for eligibility.
Groups:
- MindCotine Mobile App Program: MindCotine VR app program, a 6-week intervention to help users utilize mindfulness based skills involving virtual exposure therapy.
Period: Overall Study
Arm/Group | MindCotine Mobile App Program
Started | 20
Used the MindCotine Intervention | 9
Completed End of Treatment Survey | 8
Completed | 8
Not Completed | 12
Not completed — Withdrawal by Subject | 4
Not completed — Removed due to ineligibility | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Smoking habit [Count of Participants; unit: Participants]
  Smokes daily | 18
  Smokes some days | 2
Cigarette use - patients who smoke every day [Mean (Standard Deviation); unit: cigarettes per day] — Population: Patients who smoke every day
  cigarettes per day
    number analyzed (Participants) | 18
    (all) | 14.7 (7.2)
Cigarette use - patients who smoke some days [Mean (Standard Deviation); unit: cigarettes per week] — Population: Patients who smoke some days
  cigarettes per week
    number analyzed (Participants) | 2
    (all) | 25 (7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Registered With the MindCotine Application
Description: Total number of patients who registered with the app, out of total number of participants who were enrolled (eligible and willing to accept help with quitting). This measure is to assess whether MindCotine is a feasible smoking cessation option among patients who smoke cigarettes.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 20
Participants | 9

2. Primary Outcome: Number of Patients With Interest in the MindCotine Application
Description: Total number of patients who expressed interest in the app, out of total number of participants who were screened for enrollment. This measure is to assess whether MindCotine is a feasible smoking cessation option among patients who smoke cigarettes.
Time Frame: 6 weeks
Population: Participants who were screened for eligibility
Measure: Count of Participants; unit: Participants
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 105
Participants | 27

3. Primary Outcome: Number of Patients Who Would Recommend the MindCotine Application as a Measure of Feasibility Among Patients Who Smoke.
Description: Learning whether MindCotine is a feasible smoking cessation option among patients who smoke cigarettes.
  Interest in using the app will be calculated as total number of patients who recommend the app to others.
Time Frame: 6 weeks
Population: Participants who completed the end of treatment survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 8
Participants | 7

4. Secondary Outcome: Number of Patients Who Attempt to Quit Smoking by Using the Application
Description: Measured as the number of participants who had a 24-hour quit attempt in the past 6-weeks prior to end of treatment survey
Time Frame: 6 weeks prior to end of treatment survey
Population: Participants who completed the end of treatment survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 8
Participants | 4

5. Secondary Outcome: Number of Patients Using Cessation Medication by End of Treatment
Description: Number of participants using cessation medications among those who completed the end of treatment survey.
Time Frame: 6 weeks
Population: Participants who completed the end of treatment survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 8
Participants | 5

6. Secondary Outcome: Number of MindCotine App Program Activities Completed
Description: Program activities include VR-MET exercises and guided mindfulness-based two-dimensional video, audio, and reflection exercises.
Time Frame: 6 weeks
Population: Participants who used the app
Measure: Mean (Standard Deviation); unit: activities
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 9
activities | 13 (20.2)

7. Secondary Outcome: Number of MindCotine App Journal Entries Completed
Description: Journal Record refers to CBT-based self-reflections.
Time Frame: 6 weeks
Population: Participants who used the app
Measure: Mean (Standard Deviation); unit: Journal entries
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 9
Journal entries | 19 (26)

8. Secondary Outcome: Number of MindCotine App Coaching Engagements Completed
Description: Coaching Engagement refers to communicating with a coach through the MindCotine mobile application.
Time Frame: 6 weeks
Population: Participants who used the app
Measure: Mean (Standard Deviation); unit: Coaching engagements
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 9
Coaching engagements | 11 (12.3)

9. Secondary Outcome: Average Change in Cigarette Use
Description: Average change in cigarette use from baseline to end of treatment among patients using the MindCotine app.
Time Frame: baseline to end of treatment, up to 6 weeks
Population: patients who used the app
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 9
cigarettes | -4.1 (8)

10. Secondary Outcome: MindCotine Dropout
Description: Number of patients who withdrew or were removed from the study.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MindCotine Mobile App Program
Number analyzed (Participants) | 20
Participants | 5

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | MindCotine Mobile App Program
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MindCotine Mobile App Program (N=20)
Disorientation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Double vision (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lighheadedness (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT05220254/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT05220254/ICF_000.pdf